CLINICAL TRIAL: NCT02858141
Title: Onco-geriatric Database of Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: ONCOGEPAN
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Neoplasms
Keywords: oncogeriatric evaluation; pancreatic cancer; Database
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data collection

SUMMARY:
This data base has been set in order to gather oncogeriatric information from elderly patients with pancreatic cancer who underwent an oncogeriatric evaluation.

ONCOGEPAN database gathers data from deux institutions (Institut Paoli-Calmettes and Assistance Publique des Hôpitaux de Marseille) involved in Marseille SIRIC (Integrated Cancer Research Site).

ELIGIBILITY:
Inclusion Criteria:

* Age>70 years
* Oncogeriatric evaluation done

Exclusion Criteria:

* Patient refusal to participate in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with pancreatic cancer who underwent an oncogeriatric evaluation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Collection of oncogeriatric data for future research studies | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Crétel, Principal Investigator — Assistance Publique des Hôpitaux de Marseille; Frédérique Rousseau, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - Institut Paoli Calmettes, Marseille, Bouches du Rhône
  - Assistance Publique des Hôpitaux de Marseille, Marseille, Bouches du Rhône